CLINICAL TRIAL: NCT06660316
Title: Prevalence and Associated Risk Factors Among Nursing Students Regarding Computer Vision Syndrome
Brief Title: Risk Factors Among Nursing Students Regarding Computer Vision Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Elsayed Zaky, Principal Investigator, Cairo University
Other Study IDs: computer vision syndrome
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Computer Vision Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nursing Students - Computer Vision Syndrome Prevalence

SUMMARY:
This study aims to evaluate the prevalence of computer vision syndrome and its associated risk factors among nursing students.

DETAILED DESCRIPTION:
In the early days of technology, personal computers revolutionized the workplace, becoming a go-to tool for boosting productivity. Today, computers are not just a staple in offices-they're in nearly every home, college, and university. With this widespread use, however, comes an unexpected side effect: a growing number of people are grappling with Computer Vision Syndrome (CVS).

Imagine this: A student, spending hours in front of a screen, finishing assignments and studying for exams. The longer the screen time, the greater the chance that eye strain, dryness, and headaches will follow. Research has shown that anyone who spends over four continuous hours staring at a screen faces an increased risk of developing CVS.

The setup matters too. A poorly positioned monitor, bad lighting, or awkward posture can make matters worse. It's not just about how long you're looking at the screen-*how* you do it plays a crucial role. Correcting the distance between you and the screen, adjusting your posture, and working in an ergonomically-friendly environment can reduce the strain on your eyes and body.

Underlying eye conditions like uncorrected refractive errors or dry eye disease can also make individuals more vulnerable to CVS. Even the type of light emitted from our screens-especially blue light-can cause discomfort. For some, it's a nagging glare; for others, it's a disrupted sleep cycle that throws off their entire rhythm.

It's surprising how just a few hours of daily computer use can lead to noticeable health problems. Computers, now indispensable to our daily routines, also bring with them the risk of significant eye discomfort. Some, for instance, experience convergence insufficiency-a condition marked by eye strain, blurred vision, headaches, and neck or shoulder pain. As screen time increases, these symptoms become more pronounced. Estimates suggest that CVS affects anywhere from 64% to 90% of computer users, with around 60 million cases globally each year, and the numbers are only climbing.

In response, the American Optometric Association offers some simple solutions. One of their key recommendations is the "20-20-20 rule": every 20 minutes, take a 20-second break to look at something 20 feet away. Small changes like using glare-reducing filters can also help, although their effectiveness varies from person to person. Specialized eyewear, like blue-light blocking lenses, has shown promise in minimizing CVS symptoms.

CVS is a complex issue in our increasingly digital world. Although there's a general agreement on the major risk factors, more research is needed to fully understand the long-term impacts and what interventions work best. But in the meantime, simple actions-like making ergonomic adjustments, taking regular breaks, and investing in protective eyewear-can make a big difference. As our reliance on digital devices grows, so does the need for greater awareness and preventive measures to protect our eyes and maintain our overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Nursing Student in Collegue of Nursing - Jouf University

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any students with musculoskeletal or eye problems, unwilling to participate
Sampling Method: Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Nursing Students - Computer Vision Syndrome Prevalence | 1 month

REFERENCES:
- [Background] Mrayyan MT, Alseid ARH, Ghoolah TS, Al-Shaikh Ali MH, Mrayan M. Investigating the Prevalence of Computer Vision Syndrome (CVS) Among Undergraduate Nursing Students: A Cross-Sectional Study. SAGE Open Nurs. 2023 Aug 2;9:23779608231191883. doi: 10.1177/23779608231191883. eCollection 2023 Jan-Dec. PMID 37546525
- [Background] AlDarrab A, Khojah AA, Al-Ghazwi MH, Al-Haqbani YJ, Al-Qahtani NM, Al-Ajmi MN, Alenezi SH, Almasoud MK, Al-Yahya AF. Magnitude and Determinants of Computer Vision Syndrome among College Students at a Saudi University. Middle East Afr J Ophthalmol. 2022 Apr 30;28(4):252-256. doi: 10.4103/meajo.meajo_272_21. eCollection 2021 Oct-Dec. PMID 35719284